CLINICAL TRIAL: NCT06673342
Title: Effectiveness of a Nutritional Counseling Tool in Reducing the Amount and Frequency of Sugar Intake: A Pilot Clinical Trial
Brief Title: Effectiveness of a Nutritional Counseling Tool in Reducing the Amount and Frequency of Sugar Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5240464
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Dental Cavity; Caries,Dental
Keywords: Sugar Consumption; Nutritional Counselling
MeSH Terms: conditions — Dental Caries | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: A convenience sample of 100 participants will be enrolled for the study. Selection of participants will concur to a written consent primarily based on voluntary agreement. For each participant the following procedures will be performed:
  1. Record a thorough health history from each subject regarding past and present family health conditions and demographic information including demographic information, including age, gender, and race/ethnicity.
  2. For the control group an oral examination to visually assess the DMFT scores will be performed and added sugar consumption will be calculated using the online application, "Sugar Intake Calculator", with no additional nutritional counseling tool utilized.
  3. For the intervention group, an oral examination to visually assess the DMFT scores will be performed and added sugar consumption will be calculated using the online application, "Sugar Intake Calculator", with the intervention of Stephan's curve as a nutritional tool.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Visual assessment of DMFT, added sugar consumption calculation, frequency of snacking calculation.
- Intervention (Experimental): Visual assessment of DMFT, added sugar consumption calculation, frequency of snacking calculation, plus Stephan's Curve-based nutritional counseling.
  Interventions: Behavioral: Nutritional Counseling

INTERVENTIONS:
Behavioral: Nutritional Counseling — Nutritional counseling based on Stephan's Curve. The Stephan's curve is a diagram that shows how the acidity of the oral cavity changes with consumption of food, specifically with added sugar. A laminated Stephan's curve will be used to show the drop of pH (acidity) based on the subject's reported daily consumption of food and snacks. Recommendations will be provided on a balanced diet according to the American Dental Association guidelines and recommendations on reducing the frequency of snacking.
  Other Names: Stephan's Curve
  Arms: Intervention

SUMMARY:
The purpose of the study is to assess the effectiveness of nutritional counselling on added sugar consumption, frequency of snacking and caries experiences expressed as Decayed, Missing, and Filled Teeth score (DMFT).

DETAILED DESCRIPTION:
The study involves two visits: the first lasting approximately 30-45 minutes, and the second about 15 minutes that occurs 2 weeks after the first visit.

Procedures and Activities. Subjects will be assigned to either the control or intervention group by the toss of a coin. Subjects will provide information about their personal health history, including age, gender, and race/ethnicity. Subjects will undergo an oral examination to assess dental health through a DMFT score, which measures decayed, missing, and filled teeth. Additionally, the daily added sugar consumption will be calculated using an app called "Sugar Intake calculator." For the control group, no further nutritional advice will be given, while participants in the intervention group will receive additional guidance on sugar consumption using a tool called Stephan's curve. A log will be given to the subjects to track their daily snacking frequency and what type and amount of snack it entailed. After two weeks, subjects will return for a follow-up to evaluate any changes in dental health, sugar consumption, and snacking habits.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are 18 years or older
* Subjects who will comply with study protocol
* Subjects who can read and speak English
* Subjects available during the study period

Exclusion Criteria:

* Subjects under the age of 18
* Subjects have less than 20 teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in snacking frequency between baseline and 2 weeks | Time frame is two weeks: from baseline to the 2 weeks follow-up visit
  Subjects will self-report the snacking frequency per day at baseline and at 2 weeks. Snacking is defined as any food intake besides breakfast, lunch and dinner.
Change in amount of added sugar consumption during snacking between baseline and 2 weeks. | Time frame is two weeks: from baseline to the 2 weeks follow-up visit
  Added sugar consumption will be calculated using the "Sugar intake calculator" app at baseline and at 2 weeks follow-up. The sugar intake calculator is a free app that can generate the amount of added sugar in snacks, providing the amount in grams. Subjects will self-report the snacks that they have been consuming. The added sugar threshold for cavities is set at 40 gram/day.

SECONDARY OUTCOMES:
Change in DMFT score between baseline two weeks | Time frame is two weeks: from baseline to the 2 weeks follow-up visit
  Caries experiences is expressed as Decayed, Missing, Filled teeth and can range from 0 to 28. The higher the score the higher the caries experiences. The study investigators are going visually examine subjects' teeth and determine the DMFT score.

CONTACTS AND LOCATIONS:
Overall Officials: So Ran Kwon, DDS, MS, PhD, MS, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No